CLINICAL TRIAL: NCT01046734
Title: Virus Shedding and Environmental Deposition of Novel A(H1N1) Pandemic Influenza Virus
Brief Title: Virus Shedding and Environmental Deposition of a Novel Influenza Virus
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 09061
Record Dates: First submitted 2010-01-11; First posted 2010-01-12 (Estimated); Last update posted 2012-09-27 (Estimated); Status verified 2012-09

CONDITIONS: Novel (H1N1) Influenza
Keywords: Influenza; virus shedding; infection control; swine flu
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Adult Community
- Adult Hospital
- Children Hospital
- Children Community

SUMMARY:
An influenza pandemic has recently been declared, involving the novel A(H1N1) 'swine flu' virus. This has spread to almost 100 countries worldwide in less than two months, causing widespread disease so far in Mexico, USA and Canada. It is highly likely that over the next 12 months, many countries including the UK will be affected by widespread illness. In the UK this wave of intense flu activity is most likely to occur in late autumn 2009.

Very little is known about the new H1N1 pandemic virus. For example we do not know how long the virus is excreted by infected humans and how much virus is spread to surfaces and carried in the air. This is very important to know as soon as possible because it affects the advice that will be given to healthcare workers about controlling the spread of infection to themselves and other patients. Similarly we need this information so we can give good quality advice to families who will have to look after each other in their own homes.

The best way to obtain this information is to ask patients who get pandemic flu soon (in August, September and October) to help us by agreeing to give a daily nose swab sample for just over one week so we can see how much virus is in the nose day by day and how quickly this disappears. At the same time we will take samples from hard surfaces in a patient's room or home and sample the air using a special filter device. We can then work out how much virus is being excreted, how long the 'danger period' is, whether surfaces are more or less important than the air that we breathe (in terms of catching the virus) and if we can advise on a 'safe distance' from the patient, beyond which there is relatively little chance of catching the illness.

ELIGIBILITY:
Inclusion Criteria:

* Subject fulfils case definition
* Informed consent obtained (from Parent/Guardian where appropriate)
* Age >1 month
* Near-patient test positive for influenza A or other substantive test positive for influenza A (including 'swine flu')
* Willing to participate and agrees to allow both nasal and environmental samples to be taken

Exclusion Criteria:

* Illness for >48h (community cases)
* Illness for >96h (hospital cases)
* Existing case of ILI in the household
* A negative for swine flu (as part of NHS care)
* Has taken part in influenza research involving an investigational medicinal product within the last 3 months

Min Age: 1 Month | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adults and children with swine flu whi have had symptoms for less than 3 days
Sampling Method: Non-Probability Sample
Enrollment: 105 (Actual)
Dates: Start 2009-09; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Virus shedding and deposition as measured by virus culture and quantitative polymerase chain reaction (PCR). | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan Van-Tam, MD, Principal Investigator — University of Nottingham
Locations (3):
- United Kingdom (3):
  - Leicester University Hospitals NHS Trust, Leicester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Sheffield Teaching Hospitals NHS Trust, Sheffield